CLINICAL TRIAL: NCT02384434
Title: Utilization of Low Level Laser Therapy for Radiation Induced Dermatitis in Patients With Head and Neck Squamous Cell Carcinoma
Brief Title: Low Level Laser Therapy for Radiation Induced Dermatitis in H & N Squamous Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heath Skinner (Other)
Responsible Party: Sponsor-Investigator, Heath Skinner, Radiation Oncologist, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HCC 18-128
Record Dates: First submitted 2015-02-26; First posted 2015-03-10 (Estimated); Results first posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Low Level Laser Therapy (Other): Non-invasive, cold laser output treatment.
  Interventions: Device: THOR Laser System for Low Level Laser Therapy (LLLT)

INTERVENTIONS:
Device: THOR Laser System for Low Level Laser Therapy (LLLT) — Non-invasive, a cold laser output treatment.

SUMMARY:
This study will assess the efficacy of LLLT to mitigate and ameliorate the acneiform-rash, radiation dermatitis, and pain, while assessing its impact on patient reported quality of life.

DETAILED DESCRIPTION:
This single-arm phase I/II study establishes the safety and efficacy of low level laser therapy (LLLT) in order to mitigate radiation-induced dermatitis in patients underoing radiation therapy for head and neck squamous cell carcinoma (HNSCC). Additional objectives include assessment of patient-reported quality of life data, pain parameters and dermatologic quality of life responses. The target population is patients with histologically proven squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx who are candidates for either definitive or adjuvant therapy consisting of a chemotherapy regimen and concurrent radiation therapy.

Patients are required to have a favorable performance status (KPS greater than or equal to 70), have had no prior head and neck radiotherapy and be at least 18 years of age and able to provide consent. While receiving radiotherapy and a concurrent systemic regimen, patients will receive LLLT using a 69 diode probe with dual 660 nm and 850 nm wavelengths to at least nine treatment sites in the head and neck region for a duration of 60 seconds to each site. LLLT will be given three times in a week prior to, daily during the first week of, and at least twice weekly thereafter during radiotherapy.

Information collected includes toxicity scoring and quality of life surveys. A retrospective matched-pair design will be used to assess the rate of grade III complications compared to patients treated previously without LLLT support, with an anticipated 20% reduction in the risk of grade III dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Karnofsky performance status > 70
* Histologic proof of squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx
* No prior radiotherapy to the head and neck region.
* No previous systemic chemotherapy or targeted therapy
* Must be aware of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the nature of the therapy, alternatives, potential benefits, side-effects, risks and discomforts.
* Patients using standard therapies for cetuximab-induced acne-form rash will be included.

Exclusion Criteria:

* Evidence of distant metastasis on upright chest x-ray (CXR), computed tomography (CT) or other staging studies
* Any co-morbidity or condition of sufficient severity to limit full compliance with the protocol per assessment by the investigator
* Concurrent serious infection
* Continued use of Niacin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heath Skinner, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center - Shadyside Radiation Oncology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Level Laser Therapy
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.62 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Grade 3 or Higher Adverse Events
Description: Number of patients with documented Grade 3 or higher Adverse Events as per CTCAE v4.0.
Time Frame: Up to 12 months
Population: Patients who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 9
Participants | 9

2. Secondary Outcome: University of Washington Quality of Life Questionnaire (UW-QOL)
Description: The University of Washington Quality of Life Questionnaire (UW-QOL) consists of 12 single question domains focusing on patient health/quality of life within the past 7 days. Domains are scaled evenly from 0 (worst) to 100 (best) per the hierarchy of response. The domains are pain, appearance, activity, recreation, swallowing, chewing, speech, shoulder, taste, saliva, mood and anxiety; patient choice of up to three of these domains that have been the most important to them. There are also three global questions, one about how the patient feel relative to before they developed their cancer, one about their health-related QOL and one about overall QOL. Patients are asked to consider not only physical & mental health, but also many other factors, such as family, friends, spirituality or personal leisure activities that were important to their enjoyment of life in overall quality of life. Scores for each of the individual response options are summed to determine the domain score.
Time Frame: At Baseline
Population: Treated patients who completed UW-QOL assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 16
score on a scale
  Activity | 43.8 (21.4)
  Anxiety: number analyzed (Participants) | 15
  Anxiety | 47.3 (32.0)
  Appearance | 28.1 (25.6)
  Chewing | 40.6 (27.2)
  Mood | 35.9 (30.2)
  Pain | 48.4 (34.7)
  Recreation | 35.9 (22.3)
  Saliva: number analyzed (Participants) | 15
  Saliva | 21.3 (24.5)
  Shoulder | 21.2 (30.7)
  Speech | 15.0 (15.5)
  Swallowing | 30.0 (29.0)
  Taste | 27.5 (35.9)
  Global severity - QOL last 7 days: number analyzed (Participants) | 14
  Global severity - QOL last 7 days | 42.9 (20.5)
  Global severity - QOL since 1 mo. before cancer: number analyzed (Participants) | 15
  Global severity - QOL since 1 mo. before cancer | 31.7 (30.6)
  Overall QOL: number analyzed (Participants) | 14
  Overall QOL | 37.1 (17.3)

3. Secondary Outcome: University of Washington Quality of Life Questionnaire (UW-QOL)
Description: as for outcome 2
Time Frame: Up to 4.5 months
Population: Treated patients who completed UW-QOL assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 15
score on a scale
  Activity | 54.4 (12.1)
  Anxiety | 44.1 (29.7)
  Appearance | 35 (19.7)
  Chewing | 44.4 (34.6)
  Mood | 44.7 (28.3)
  Pain | 49.4 (26.7)
  Recreation | 49.4 (20)
  Saliva | 51.8 (25.7)
  Shoulder | 20.3 (29.4)
  Speech | 27.3 (29.1)
  Swallowing | 41.6 (29.1)
  Taste | 79.8 (25)
  Global severity - QOL last 7 days | 55.3 (18.1)
  Global severity - QOL since 1 mo. before cancer | 51.4 (19.3)
  Global severity - Overall QOL | 50.7 (21.7)

4. Secondary Outcome: University of Washington Quality of Life Questionnaire (UW-QOL)
Description: as for outcome 2
Time Frame: 4.5-7.5 months
Population: Treated patients who completed UW-QOL assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 8
score on a scale
  Activity | 43.8 (17.7)
  Anxiety: number analyzed (Participants) | 7
  Anxiety | 47.1 (21.4)
  Appearance | 25.0 (18.9)
  Chewing: number analyzed (Participants) | 7
  Chewing | 32.1 (31.3)
  Mood: number analyzed (Participants) | 7
  Mood | 35.7 (24.4)
  Pain | 34.4 (26.5)
  Recreation: number analyzed (Participants) | 7
  Recreation | 39.3 (19.7)
  Saliva: number analyzed (Participants) | 7
  Saliva | 48.6 (28.5)
  Shoulder: number analyzed (Participants) | 7
  Shoulder | 30.7 (29.5)
  Speech: number analyzed (Participants) | 7
  Speech | 8.6 (14.6)
  Swallowing: number analyzed (Participants) | 7
  Swallowing | 31.4 (33.4)
  Taste: number analyzed (Participants) | 7
  Taste | 52.9 (21.4)
  Global severity - QOL last 7 days: number analyzed (Participants) | 7
  Global severity - QOL last 7 days | 51.4 (10.7)
  Global severity - QOL since 1 mo. before cancer: number analyzed (Participants) | 7
  Global severity - QOL since 1 mo. before cancer | 28.6 (26.7)
  Global severity - Overall QOL: number analyzed (Participants) | 7
  Global severity - Overall QOL | 42.9 (13.8)

5. Secondary Outcome: University of Washington Quality of Life Questionnaire (UW-QOL)
Description: as for outcome 2
Time Frame: 7.5-10.5 months
Population: Treated patients who completed UW-QOL assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 7
score on a scale
  Activity | 46.4 (22.5)
  Anxiety | 37.9 (24.8)
  Appearance | 21.4 (18.7)
  Chewing | 25 (25)
  Mood | 50 (25)
  Pain | 30.4 (26.9)
  Recreation | 41.1 (23.6)
  Saliva | 28.6 (31.3)
  Shoulder | 14.3 (27)
  Speech | 18.6 (26.7)
  Swallowing | 15.7 (15.9)
  Taste | 49.3 (28.1)
  Global severity - QOL last 7 days: number analyzed (Participants) | 6
  Global severity - QOL last 7 days | 46.7 (15.1)
  Global severity - QOL since 1 mo. before cancer: number analyzed (Participants) | 6
  Global severity - QOL since 1 mo. before cancer | 16.7 (21.9)
  Global severity - Overall QOL: number analyzed (Participants) | 6
  Global severity - Overall QOL | 45.0 (15.2)

6. Secondary Outcome: University of Washington Quality of Life Questionnaire (UW-QOL)
Description: as for outcome 2
Time Frame: 10.5-13.5 months
Population: Treated patients who completed UW-QOL assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 4
score on a scale
  Activity | 37.5 (14.4)
  Anxiety | 17.5 (35.0)
  Appearance | 12.5 (14.4)
  Chewing | 12.5 (25)
  Mood | 18.8 (12.5)
  Pain | 28.1 (32.9)
  Recreation | 43.8 (12.5)
  Saliva | 25.0 (33.2)
  Shoulder | 30 (35.6)
  Speech | 3.8 (7.5)
  Swallowing | 15 (17.3)
  Taste | 27.5 (20.6)
  Global severity - QOL last 7 days | 42.5 (5)
  Global severity - QOL since 1 mo. before cancer | 21.9 (21.3)
  Global severity - Overall QOL | 30 (11.5)

7. Secondary Outcome: University of Washington Quality of Life Questionnaire (UW-QOL)
Description: as for outcome 2
Time Frame: 13.5-16.5 months
Population: Treated patients who completed UW-QOL assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 4
score on a scale
  Activity | 46.9 (29.5)
  Anxiety | 12.5 (25)
  Appearance | 6.2 (12.5)
  Chewing | 12.5 (25)
  Mood | 18.8 (23.9)
  Pain | 0 (0)
  Recreation | 43.8 (31.5)
  Saliva | 7.5 (15.0)
  Shoulder | 17.5 (35)
  Speech | 7.5 (15)
  Swallowing | 25.0 (33.2)
  Taste | 22.5 (15)
  Global severity - QOL last 7 days | 45 (10)
  Global severity - QOL since 1 mo. before cancer | 50 (20.4)
  Global severity - Overall QOL | 35 (19.1)

8. Secondary Outcome: University of Washington Quality of Life Questionnaire (UW-QOL)
Description: as for outcome 2
Time Frame: after 16.5 months, up to 48.9 months
Population: Treated patients who completed UW-QOL assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 4
score on a scale
  Activity | 35.4 (12.5)
  Anxiety | 21 (31.5)
  Appearance | 11.6 (13.5)
  Chewing | 16.7 (23.6)
  Mood | 25.6 (29.2)
  Pain | 17.6 (32.8)
  Recreation | 40.8 (16.6)
  Saliva | 15 (17.3)
  Shoulder | 14 (16.8)
  Speech | 2.5 (5.0)
  Swallowing | 33.9 (45.3)
  Taste | 19. (9.6)
  Global severity - QOL last 7 days | 46.8 (10.4)
  Global severity - QOL since 1 mo. before cancer | 38.8 (27.1)
  Global severity - Overall QOL | 40.4 (13.8)

9. Secondary Outcome: Brief Pain Inventory (BPI)
Description: Pain parameters assessed using Brief Pain Inventory (BPI). The BPI allows patients to rate the severity of their pain and the degree to which their pain interferes (impact on) with common dimensions of feeling and function. No scoring algorithm, but "worst pain" or the arithmetic mean of the four severity items (Pain Worst in last week, Pain least in last week, Average Pain, Pain right now) indicates pain severity; the arithmetic mean of the seven interference items (General Activity, Mood, Walking Ability, Normal Work, Relationships, Sleep, Enjoyment of Life) measures how much pain impacted/interfered with a patient's various daily activities. Total scores range = 0 -10 for each item (mean of patient scores for each item).
  Pain and interference of pain in daily activities is scored as follows: 1 - 4 = Mild, 5 - 6 = Moderate, 7 - 10 = Severe
  Higher scores indicate greater pain and/or greater impact of pain and interference in activity, per item.
Time Frame: Baseline
Population: Treated patients who completed BPI assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 15
score on a scale
  General Activity | 6.3 (2.6)
  Enjoyment of Life | 5.8 (2.8)
  Mood | 5.0 (3.1)
  Normal Work | 5.6 (3.3)
  Relationships | 4.3 (3.7)
  Sleep | 6.3 (2.7)
  Walking Ability: number analyzed (Participants) | 14
  Walking Ability | 3.0 (3.8)
  Average pain | 5.5 (2.1)
  Pain least in last week | 4.0 (2.8)
  Pain right now | 4.8 (2.9)
  Pain Worst in last week | 7.1 (2.2)

10. Secondary Outcome: Brief Pain Inventory (BPI)
Description: as for outcome 9
Time Frame: Up to 4.5 months
Population: Treated patients who completed BPI assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 11
score on a scale
  General Activity: number analyzed (Participants) | 10
  General Activity | 5.5 (2.6)
  Enjoyment of Life: number analyzed (Participants) | 9
  Enjoyment of Life | 5.1 (3.4)
  Mood: number analyzed (Participants) | 10
  Mood | 5.2 (3.4)
  Normal Work: number analyzed (Participants) | 10
  Normal Work | 3.7 (3.1)
  Relationships: number analyzed (Participants) | 10
  Relationships | 3.6 (2.8)
  Sleep: number analyzed (Participants) | 10
  Sleep | 5.9 (3.1)
  Walking Ability: number analyzed (Participants) | 10
  Walking Ability | 3.3 (3.2)
  Average pain | 5 (2.7)
  Pain least in last week | 4.1 (2.3)
  Pain right now: number analyzed (Participants) | 10
  Pain right now | 5.4 (3.2)
  Pain Worst in last week | 6.3 (3.3)

11. Secondary Outcome: Brief Pain Inventory (BPI)
Description: as for outcome 9
Time Frame: 4.5-7.5 months
Population: Treated patients who completed BPI assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 3
score on a scale
  General Activity | 2.7 (3.8)
  Mood | 4.0 (4.0)
  Walking Ability | 4.3 (4.5)
  Normal Work | 4.3 (3.5)
  Relationships | 3.7 (3.8)
  Sleep | 4.3 (3.5)
  Enjoyment of Life | 4.3 (3.5)
  Pain Worst in last week | 5.8 (3.5)
  Pain least in last week (N | 3.5 (3.4)
  Average pain | 4.8 (2.2)
  Pain right now | 4.3 (3.3)

12. Secondary Outcome: Brief Pain Inventory (BPI)
Description: as for outcome 9
Time Frame: 7.5-10.5 months
Population: Treated patients who completed BPI assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 4
score on a scale
  General Activity | 3 (2.4)
  Enjoyment of Life | 5.2 (1.7)
  Mood | 2.6 (2.1)
  Normal Work | 2.5 (2.9)
  Relationships | 0.8 (1.5)
  Sleep | 5.1 (3)
  Walking Ability | 3.5 (3.1)
  Average pain | 3.8 (2.8)
  Pain least in last week | 3.1 (2.9)
  Pain right now | 3.9 (3.4)
  Pain Worst in last week | 4.8 (2.4)

13. Secondary Outcome: Brief Pain Inventory (BPI)
Description: as for outcome 9
Time Frame: 10.5-13.5 months
Population: Treated patients who completed BPI assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 2
score on a scale
  General Activity | 0.5 (0.7)
  Enjoyment of Life | 1.5 (2.1)
  Mood | 0.5 (0.7)
  Normal Work | 0.5 (0.7)
  Relationships | 0.0 (0.0)
  Sleep | 3.0 (4.2)
  Walking Ability | 0.5 (0.7)
  Average pain | 3.5 (3.5)
  Pain least in last week | 3.0 (4.2)
  Pain right now | 3.0 (4.2)
  Pain Worst in last week | 4.0 (2.8)

14. Secondary Outcome: Brief Pain Inventory (BPI)
Description: as for outcome 9
Time Frame: 13.5-16.5 months
Population: Treated patients who completed BPI assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 2
score on a scale
  General Activity | 6.5 (3.5)
  Enjoyment of Life | 6.5 (4.9)
  Mood | 6.5 (3.5)
  Normal Work | 7.0 (2.8)
  Relationships | 4.5 (4.9)
  Sleep | 6.5 (4.9)
  Walking Ability | 4.5 (6.4)
  Average pain | 4.5 (4.9)
  Pain least in last week | 5.0 (4.2)
  Pain right now | 5.0 (7.1)
  Pain Worst in last week | 5.5 (6.4)

15. Secondary Outcome: Brief Pain Inventory (BPI)
Description: as for outcome 9
Time Frame: after 16.5 months, up to 48.9 months
Population: Treated patients who completed BPI assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 4
score on a scale
  General Activity | 2.2 (2.9)
  Enjoyment of Life | 2 (2.4)
  Mood | 1.8 (2.6)
  Normal Work | 2.4 (2.9)
  Relationships | 1.2 (1.5)
  Sleep | 1.7 (2.8)
  Walking Ability | 2.5 (3.1)
  Average pain | 2 (2.6)
  Pain least in last week | 1.5 (2.1)
  Pain right now | 1.7 (3.1)
  Pain Worst in last week | 2.4 (3.0)

16. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: Dermatologic quality of life responses measured using the Dermatology Life Quality Index (DLQI). The DLQI is a ten-question questionnaire designed to measure the health-related quality of life of adult patients suffering from a skin disease, the impact of the skin disease on the patient's life over the previous week. Each question is scored from 0 to 3, giving a possible score range from 0 (meaning no impact on quality of life) to 30 (meaning maximum impact on quality of life). Scoring bands: 0-1 = No effect on patient's life, 2-5 = Small effect, 6-10 = Moderate effect, 11-20 = Very large effect, 21-30 = Extremely large effect. Higher scores indicate greater impact of skin disease on patient's life.
Time Frame: Baseline
Population: Treated patients who completed DLQI assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 15
score on a scale
  Activity | 4.1 (0.8)
  Appearance | 3.7 (0.6)
  Clothes | 4.1 (0.6)
  Messy | 4.3 (0.6)
  Pain | 3.3 (1.0)
  Problems | 4.2 (0.6)
  Sexual | 4.1 (1.0)
  Social | 4.1 (0.8)
  Sport | 4.1 (1.0)
  Studying | 1.3 (1.5)
  Working | 2.5 (0.5)

17. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: as for outcome 16
Time Frame: Up to 4.5 months
Population: Treated patients who completed DLQI assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 14
score on a scale
  Activity | 3.3 (1.2)
  Appearance | 3.2 (0.9)
  Clothes | 3.2 (1.0)
  Messy | 3.4 (0.7)
  Pain | 2.6 (0.9)
  Problems | 3.7 (0.6)
  Sexual | 4.0 (0.9)
  Social | 3.3 (1)
  Sport | 4.2 (1)
  Studying | 0.6 (0.9)
  Working | 2.7 (0.3)

18. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: as for outcome 16
Time Frame: 4.5 - 7.5 months
Population: Treated patients who completed DLQI assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 4
score on a scale
  Activity | 3.8 (0.5)
  Appearance | 3.5 (0.6)
  Clothes | 4.2 (0.5)
  Messy | 4.0 (0.8)
  Pain | 3.5 (0.6)
  Problems | 4.5 (0.6)
  Sexual | 4.0 (0.8)
  Social | 3.8 (0.5)
  Sport | 4.2 (1.0)
  Studying | 0.8 (1.5)
  Working | 2.8 (0.5)

19. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: as for outcome 16
Time Frame: 7.5-10.5 months
Population: Treated patients who completed DLQI assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 8
score on a scale
  Activity | 3.8 (0.5)
  Appearance | 3.8 (0.5)
  Clothes | 3.9 (0.4)
  Messy | 4.1 (0.6)
  Pain | 3.3 (0.8)
  Problems | 3.8 (0.5)
  Sexual | 3.9 (0.9)
  Social | 3.9 (0.6)
  Sport | 3.5 (1.3)
  Studying | 2.4 (1.1)
  Working | 1.9 (0.4)

20. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: as for outcome 16
Time Frame: 10.5-13.5 months
Population: Treated patients who completed DLQI assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 4
score on a scale
  Activity | 4.2 (0.5)
  Appearance | 4.0 (0.0)
  Clothes | 4.0 (0.6)
  Messy | 4.0 (0.6)
  Pain | 3.5 (1)
  Problems | 4.2 (0.5)
  Sexual | 4.2 (0.5)
  Social | 4.2 (0.5)
  Sport | 4.4 (0.5)
  Studying | 1.9 (1.4)
  Working | 2.4 (0.5)

21. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: as for outcome 16
Time Frame: 13.5-16.5 months
Population: Treated patients who completed DLQI assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 4
score on a scale
  Activity | 4.2 (0.5)
  Appearance | 4.0 (0.0)
  Clothes | 4.0 (0.0)
  Messy | 4.2 (0.5)
  Pain | 3.8 (0.5)
  Problems | 4.0 (0.0)
  Sexual | 4.5 (0.6)
  Social | 4.2 (0.5)
  Sport | 4.0 (0.8)
  Studying | 2.2 (1.5)
  Working | 2.2 (0.5)

22. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: as for outcome 16
Time Frame: after 16.5 months, up to 48.9 months
Population: Treated patients who completed DLQI assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 4
score on a scale
  Activity | 3.8 (0.5)
  Appearance | 4 (0.1)
  Clothes | 4 (0.1)
  Messy | 4.3 (0.5)
  Pain | 3.5 (0.5)
  Problems | 4 (0.1)
  Sexual | 4.3 (0.5)
  Social | 4 (0.1)
  Sport | 4.1 (0.1)
  Studying | 2.2 (1.4)
  Working | 2.3 (0.5)

ADVERSE EVENTS:
Time Frame: Up to 5 years and 5.5 months for the study population.
Arm/Group | Low Level Laser Therapy
All-Cause Mortality (participants affected / at risk) | 12/16
Serious Adverse Events (participants affected / at risk) | 9/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Level Laser Therapy (N=16)
Dysphagia (Gastrointestinal disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 1
Pain (General disorders) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Level Laser Therapy (N=16)
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 12
Dysphagia (Gastrointestinal disorders) | 12
Esophagitis (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 15
Pain (General disorders) | 15
Dermatitis radiation (Injury, poisoning and procedural complications) | 12
Weight loss (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 11
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 11
Headache (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT02384434/Prot_SAP_000.pdf